CLINICAL TRIAL: NCT05045040
Title: Effectiveness of a Facilitating Program Utilizing a Mobile Application for Initiating Advanced Care Planning Discussions Between Patients with Advanced Cancer and Healthcare Providers: Protocol for a Randomized Controlled Trial (J-SUPPORT 2104)
Brief Title: Empathetic Communication Facilitation Program for Early Initiation of End-of-life Discussions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yosuke Uchitomi (Other Government)
Responsible Party: Sponsor-Investigator, Yosuke Uchitomi, Chief of Innovation Center for Supportive, Palliative and Psychosocial Care, National Cancer Center Hospital, National Cancer Center, Japan
Organization: National Cancer Center, Japan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: J-SUPPORT2104; 20EA1010 (Other Grant/Funding Number: Health and Labor Sciences Research Grants)
Record Dates: First submitted 2021-08-24; First posted 2021-09-16 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: End of Life Care; Advanced Cancer; Recurrent Cancer
Keywords: Advance Care Planning; Communication; Decision Making; Neoplasms; Palliative Care
MeSH Terms: conditions — Recurrence; Communication; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobile-based empathetic communication support program group (Experimental): Patients are provided a mobile-based empathetic communication support program to promote ACP discussion for patients with advanced cancer and physicians. The experimental group also receives the usual care as is standard practice.
  Interventions: Behavioral: Mobile-based empathetic communication support program to promote ACP discussion
- Usual care group (No Intervention): Patients receive the usual care. The usual care includes routine medical treatment and care by physicians, nurses, pharmacists, and others as well as support from the palliative care team and others as per the patient's situation.

INTERVENTIONS:
Behavioral: Mobile-based empathetic communication support program to promote ACP discussion — Patients in the intervention group are provided a mobile-based empathic communication support program-an app on a mobile phone. The app comprises a QPL (46 questions in eight categories) and questions about the patient's preferred treatment and end-of-life care based on their values and goals. Then, they proceed with the content themselves, at home or anywhere, at any time. Between app registration and the next outpatient visit, the patient is interviewed (by phone or in person) by a nurse or a clinical psychologist, who helps them prepare for the discussion with the physician and asks questions based on the patient's app responses for 30 minutes to an hour. During the outpatient visit, feedback is provided to patients and their physicians based on the interview. The duration between the start of app use and the next consultation is a minimum of one week and a maximum of four weeks.
  Arms: Mobile-based empathetic communication support program group

SUMMARY:
Background: The National Comprehensive Cancer Network Clinical Practice Guidelines in Oncology: palliative care recommends discussing advance care planning (ACP) when patients' estimated life expectancy is reduced from a year to months. Discussions about ACP focus on communication among patients, their caregivers, and healthcare providers to achieve cancer-related treatment and care consistent with the patient's preferences based on their values and goals. ACP can improve outcomes for patients and caregivers; however, provision of ACP to patients remain low. This may be because of the complexity of ACP in clinical practice.

A Question Prompt List (QPL) is a structured question list encouraging patients to put forward their queries to physicians and promote discussion between patients and physicians during medical consultations. Our preliminary study found that for patients with advanced cancer after standard chemotherapy, face-to-face interventions by nurses or clinical psychologists using a QPL about treatment and care, which is consistent with the patient's preferences based on their values and goals promoted empathetic communication between patients and their physicians. In recent years, however, ensuring adequate time during outpatient visits has become difficult due to increased numbers of outpatients and shortages of corresponding medical personnel. Therefore, intervention methods not restricted by location or time are needed. Thus, the investigators develop a mobile-based empathetic communication support program, including a QPL, to facilitate discussions about patients' values and goals with their physicians.

Purpose: This study examines whether a mobile-based empathetic communication support program, which intends to promote ACP discussions in earlier stages of advanced cancer treatment, improves such communication behaviors of patients with advanced cancer and their physicians.

Main contents of the intervention: Patients in the intervention group are provided a mobile-based empathetic communication support program-a mobile application (app). The app comprises a QPL (46 questions in eight categories) and questions about the patient's preferred treatment and end-of-life care based on their values and goals. After registering on the app, patients are first given a program overview and instructions for using the app. Then, they proceed with the content themselves, at home or anywhere else, at any time. Between app registration and the next outpatient visit, the patient is interviewed (by phone or in person) by a nurse or a clinical psychologist, who helps them prepare for the discussion with the physician and asks questions based on the patient's app responses for 30 minutes to an hour. During the outpatient visit, patients and their physicians are provided feedback based on the interview.

Study participants: Overall, 264 patients with advanced or recurrent cancer are recruited from four departments (respiratory medicine, gastroenterology, hepatobiliary medicine, and oncology) in the outpatient clinic of the National Cancer Center Hospital, Japan.

Outcome measurement: The primary outcome of this trial is the Reassurance and Emotional support score of physician behavior measured using the SHARE model at the first visit after the intervention. SHARE is a conceptual communication skills model comprising 26 items and four subscales, categorized as S: Supportive environment, H: How to deliver bad news, A: Additional information, and RE: Reassurance and Emotional support. Reassurance and Emotional support assesses physicians' behavior in providing reassurance and addressing patients' emotions with empathetic responses (e.g., remaining silent out of concern for patient's feelings or accepting patient's expression of emotions). The conversation between patients and the physicians is audio-recorded, and a third person's impression of the physician's communication behavior during the outpatient consultation is scored on a 5-point scale from 0: not applicable at all to 4: strongly applicable. Scoring will be conducted by multiple raters blinded to the assignment. Raters are trained in conversation analysis with a manual, and inter- and intra-rater agreements will be checked in advance.

Secondary outcomes are as follows: 1) the patient-physician behavioral assessment based on the conversation analysis manual, 2) number of conversations about ACP, 3) psychological distress, 4) quality of life, 5) medical care use, 6) app use, 7) feasibility of intervention program, 8) patients' satisfaction of the consultation, 9) care goals, and 10) preferred place for future care. The investigators chose these outcomes for their comparability with previous studies.

DETAILED DESCRIPTION:
After obtaining written informed consent, patients who satisfy the criteria are assigned using a minimizing method to either an intervention or control group with stratification factors of the clinical department (respiratory medicine, gastroenterology, hepatobiliary medicine, and oncology), gender (male and female), and age (at age 64 years or younger/65 years or older). Within strata, patients are randomized to the intervention arm and the control arm in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable (Union for International Cancer Control, UICC stage III or IV) or recurrent cancer.
* Patients who are judged by the attending physician to meet the Surprise Question tool (Bernacki et al., 2019; Moss et al., 2010).
* Patients aged 20 years or older.
* Patients who have an ECOG Performance status 0-2.

  (0) Fully active and able to carry on all pre-disease performance without restriction. (1) Restricted in physically strenuous activity but ambulatory and able to engaged in light or sedentary work, e.g., light house or office work. (2) Ambulatory and capable of all self-care but unable to engage in any work activities; up and about more than 50% of waking hours. (3) Capable of only limited self-care; confined to a bed or chair for more than 50% of waking hours. (4) Completely disabled; cannot carry on any selfcare; completely confined to a bed or chair
* Patients who have provided written consent to participate in the study
* Patients who are able to read, write, and understand Japanese.

Exclusion Criteria:

* Patients judged by the attending physician to have a serious cognitive decline, such as delirium or dementia
* Patients with an estimated prognosis of three or fewer months
* Patients who are otherwise judged by the attending physician to be unsuitable for this study
* Patients who are in the middle of other psychological or communication support protocol interventions at the time of enrollment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Oncologists' communication behaviors - RE subscale (reassurance and emotional support) from the SHARE scoring manual | The first post-baseline visit (up to 4 weeks)
  SHARE comprises 26 items and four subscales categorized as S: Supportive environment, H: How to deliver bad news, A: Additional information, and RE: Reassurance and Emotional support. The investigators focus on RE, which assesses oncologists' behavior in providing reassurance and their empathetic responses to participants' emotions. Patient-physician conversation is audio-recorded, and a third person's impression of the physician's communication behavior is scored on a five-point scale (0: not applicable at all, 4: strongly applicable). Higher score indicates better communication behavior.
  References:
  A randomized controlled trial with a cluster of oncologists evaluating of an integrated communication support program for oncologists, caregivers, and patients with rapidly progressing advanced cancer on patient-centered conversation: J-SUPPORT 1704 study. ASCO Annual Meeting; 2021. J Clin Oncol.
  Fujimori M, et al. Palliat Support Care 2014;12(5):379-86.

SECONDARY OUTCOMES:
The score of oncologists' communication behaviors - S, H, and A subscales from the SHARE scoring manual | The first post-baseline visit (up to 4 weeks)
  SHARE comprises 26 items and four subscales categorized as S: Supportive environment, H: How to deliver bad news, A: Additional information, and RE: Reassurance and Emotional support. Oncologists' communication behaviors at visit T1 are evaluated using the S, H, and A subscales of the SHARE manual. Patient-physician conversation is audio-recorded, and a third person's impression of the physician's communication behavior is scored on a five-point scale (0: not applicable at all, 4: strongly applicable). Higher score indicates better communication behavior.
Communication behaviors between participants and oncologists | The first post-baseline visit (up to 4 weeks)
  The audio-recorded conversations between the participant and oncologists are coded, and the communication behaviors are counted using a computer version of the RIAS (the Roter interaction process analysis system).
  RIAS has 42 categories for coding in-consultation communication behaviors. Two blinded, trained coders assign one of the 42 codes to each utterance of the participants and oncologists.
  The number of utterances in each cluster is also evaluated. Coders are trained and certified at the official training site, the RIAS Study Group Japan Chapter. Ten percent of the total consultations (25 consultations) are double-coded, and inter-coder reliability is examined regarding the degree of agreement for the identification of utterances and coding of each utterance. The reliability is high (0.7-0.8) in previous studies.
  References:
  Roter D, et al. Patient Educ Couns 2002;46(4):243-51. Ishikawa H, et al. Soc Sci Med 2002;55(2):301-11.
Number of ACP-related topics in the consultation | The first post-baseline visit (up to 4 weeks)
  Conversations between patients and oncologists are coded and counted based on a conversation analysis manual.
  The coders, blinded to assignment, extract the patients' questions and the cues that the patient is trying to initiate or control the conversation. Next, the coders identify and categorize the patients' questions and cues into ACP topics along with the QPL questions. The patients' questions are listed on the intervention feedback sheet given to the oncologist before the visit; therefore, the oncologist may begin to discuss the patients' questions. The following ACP-related topics are included in the QPL: future treatment, future living arrangements, when standard treatment is no longer available, prognosis for the future, and family support.
  Reference:
  Epstein RM, et al. JAMA Oncol 2017;3(1):92-100.
Psychological distress | Baseline, The first post-baseline visit (up to 4 weeks), the second post-baseline visit (up to 4 weeks from the previous visit), 12 weeks after the baseline, and 24 weeks after the baseline
  The HADS (Hospital Anxiety and Depression Scale) is a 14-item self-administered questionnaire that measures psychological distress in patients. It includes subscales for depression (7 items) and anxiety (7 items). Responses are selected from four options, and scores range from 0 to 21 for each subscale. The cut-off scores are 4/5 points on the depression scale, 7/8 points on the anxiety scale, and 10/11 points on a total score. Higher scores suggest a higher possibility of having symptoms.
  References:
  Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatrica Scandinavica 1983;67(6):361-70.
  Kugaya A, Akechi T, Okuyama T, et al. Screening for psychological distress in Japanese cancer patients. Japanese journal of clinical oncology 1998;28(5):333-38.
Quality of life measured by the EORTC-QLQ-C30 | Baseline, the second post-baseline visit (up to 4 weeks from the previous visit), 12 weeks after the baseline, and 24 weeks after the baseline
  The European Organization for Research and Treatment of Cancer, Quality of Life Questionnaire (EORTC-QLQ-C30) is an integrated system for assessing the health-related quality of life (QoL) of cancer patients. The QLQ-C30 includes functional scales, symptom scales, and a global health status/QoL scale. The scales and single-item measures have a score range of 0 to 100. A high score on the functional scale indicates high functioning, that on the global health and quality of life scale indicates high health status, whereas one on the symptom scale and financial impact indicates a high level of symptoms or problems.
  References:
  Aaronson NK, et al. J National Cancer Institute 1993;85(5):365-76. Kobayashi K, et al. Eur J Cancer 1998;34(6):810-5.
Participants' care goals | Baseline, 12 weeks after the baseline, and 24 weeks after the baseline
  Participants are asked about their care goals. The treatment options are as follows: 1) I would like to receive treatment to relieve symptoms so that I can live a peaceful life, but I do not want to receive any cancer treatment that has side effects or burden, 2) I would like to receive cancer treatment that has few side effects and low burden so that I can continue my life as before, 3) I have important things I need to do, so I would like to receive cancer treatment even if there are side effects or burden, so that I can accomplish them, 4) I would like to receive all cancer treatments, regardless of their side effects or burden, so that I can live as long as possible.
Participants' preferred places for spending their final days | Baseline, 12 weeks after the baseline, and 24 weeks after the baseline
  Participants are asked about the places where they would prefer to spend their final days.
  The options for participants' preferred place where they would spend their final days are as follows: 1) home, 2) a nearby hospital, 3) a palliative care hospital or ward, 4) the hospital where they are receiving treatment, and 5) others.
Participant satisfaction with their oncologists' consultation | The first post-baseline visit (up to 4 weeks)
  The Patient Satisfaction Survey measures patient satisfaction of the consultation; it comprises five items: needs addressed, active involvement in the interaction, information received, emotional support received, and interaction in general. Each item is rated on an 11-point scale from 0 (not satisfied at all) to 10 (very satisfied). Total satisfaction is obtained by summing the answers to the questions.
  References:
  Ong LM, et al. Patient Educ Couns 2000;41(2):145-56. Blanchard CG, et al. Cancer 1986;58(2):387-93. Zandbelt LC, et al. J Gen Intern Med 2004;19(11):1088-95.
Feasibility of the intervention | The first post-baseline visit (up to 4 weeks)
  The intervention's feasibility is evaluated according to the participants' assessment of the app's usability, the time taken for interventions, and app log records. The app's usability is determined by the following five questions: 1) Were the questions you wanted to ask identified by the time you saw your oncologist? 2) Did you understand and use the app? 3) Was the app program helpful? 4) Were you comfortable with the app program? 5) Was the telephone or in-person assistance helpful? Participants rate each item on an 11-point scale (0, not satisfied at all, to 10, very satisfied). The intervention provider records the time taken for the intervention on the intervention report form. App log records, including the time spent browsing and the operation status of the intervention program, are provided by the app developer.
Medical care utilization: the presence or absence of anticancer treatment and a reason for treatment termination if it is discontinued | 24 weeks after the baseline
  This is obtained from the electrical medical record of each participant at the 6-month follow-up. If the participant is not alive at 6 months, a medical record survey based on information at the time of death will be conducted.
Medical care utilization: unscheduled outpatient visits | 24 weeks after the baseline
  This is obtained from the electrical medical record of each participant at the 6-month follow-up. If the participant is not alive at 6 months, a medical record survey based on information at the time of death will be conducted.
Medical care utilization: hospitalization | 24 weeks after the baseline
  This is obtained from the electrical medical record of each participant at the 6-month follow-up. If the participant is not alive at 6 months, a medical record survey based on information at the time of death will be conducted.
Medical care utilization: ICU admission | 24 weeks after the baseline
  This is obtained from the electrical medical record of each participant at the 6-month follow-up. If the participant is not alive at 6 months, a medical record survey based on information at the time of death will be conducted.
Medical care utilization: use of end-of-life care consultations | 24 weeks after the baseline
  This is obtained from the electrical medical record of each participant at the 6-month follow-up. If the participant is not alive at 6 months, a medical record survey based on information at the time of death will be conducted.
Medical care utilization: use of palliative care services | 24 weeks after the baseline
  This is obtained from the electrical medical record of each participant at the 6-month follow-up. If the participant is not alive at 6 months, a medical record survey based on information at the time of death will be conducted.
Cancer type | Baseline
  This is obtained from medical records.
Length of time since diagnosis in months | Baseline
  This is obtained from medical records.
Age in years | Baseline
  This is obtained from medical records.
Sex | Baseline
  This is obtained from medical records.
Educational background | Baseline
  Participants answer the questionnaire. The options are as follows: 1) graduated junior high school, 2) graduated high school, 3) junior college or technical college, and 3) college or graduate school.
Employment | Baseline
  Participants answer the questionnaire. The options are as follows: 1) full-time worker, 2) part-time worker, 3) on left, 4) unemployed, 5) housewife/househusband, 6) retired, 7) student, and 8) others.
Financial status | Baseline
  Participants answer the questionnaire. The options are as follows: 1) enough, 2) fairly sufficient, 3) rather insufficient, 4) somewhat insufficient, and 5) insufficient.
Family member | Baseline
  Participants answer the questionnaire. The options are as follows (multiple): 1) living alone, 2) living with a spouse or partner, 3) living with children, and 4) living with a person who needs care.
Methods of hospital visits | Baseline
  Participants answer the questionnaire. The options are as follows: 1) by train, 2) by bus, 3) driving a car, and 4) by other. Whether there is a family member or other person who can accompany them.
Times of hospital visits in min | Baseline
  Participants are asked how long it usually takes to get to the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Yosuke Uchitomi, MD, PhD, Principal Investigator — National Cancer Center, Japan
Locations (1):
- National Cancer Center Hospital, National Cancer Center, Tokyo, Chuo-ku, Japan

IPD SHARING:
Plan to Share IPD: Yes
Data obtained from this study may be used for secondary purposes at the request of the submitting publisher or other researchers in a form that is not linked to personal information. The study protocol, data definition tables, and dataset will be uploaded to the UMIN-Individual Case Data Repository at https://www.umin.ac.jp/icdr/index-j.html
Supporting Information: Study Protocol
Time Frame: Prior to public release, individual requests will be handled on a case-by-case basis.
Access Criteria: Undecided
URL: https://www.umin.ac.jp/icdr/index-j.html

REFERENCES:
- [Background] Fujimori M, Shirai Y, Asai M, Akizuki N, Katsumata N, Kubota K, Uchitomi Y. Development and preliminary evaluation of communication skills training program for oncologists based on patient preferences for communicating bad news. Palliat Support Care. 2014 Oct;12(5):379-86. doi: 10.1017/S147895151300031X. Epub 2013 Nov 4. PMID 24182602
- [Background] Bernacki R, Paladino J, Neville BA, Hutchings M, Kavanagh J, Geerse OP, Lakin J, Sanders JJ, Miller K, Lipsitz S, Gawande AA, Block SD. Effect of the Serious Illness Care Program in Outpatient Oncology: A Cluster Randomized Clinical Trial. JAMA Intern Med. 2019 Jun 1;179(6):751-759. doi: 10.1001/jamainternmed.2019.0077. PMID 30870563
- [Background] Moss AH, Lunney JR, Culp S, Auber M, Kurian S, Rogers J, Dower J, Abraham J. Prognostic significance of the "surprise" question in cancer patients. J Palliat Med. 2010 Jul;13(7):837-40. doi: 10.1089/jpm.2010.0018. PMID 20636154
- [Derived] Obama K, Fujimori M, Okamura M, Kadowaki M, Ueno T, Boku N, Mori M, Akechi T, Yamaguchi T, Oyamada S, Okizaki A, Miyaji T, Sakurai N, Uchitomi Y. Effectiveness of a facilitation programme using a mobile application for initiating advance care planning discussions between patients with advanced cancer and healthcare providers: protocol for a randomised controlled trial (J-SUPPORT 2104). BMJ Open. 2023 Mar 28;13(3):e069557. doi: 10.1136/bmjopen-2022-069557. PMID 36977536